CLINICAL TRIAL: NCT04850287
Title: Improving Health Awareness Using Social Network Interventions
Acronym: SNI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1596733
Record Dates: First submitted 2021-04-07; First posted 2021-04-20 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator)
  Interventions: Behavioral: Digital Sensors for Population Awareness about Health Issues using Social Media
- Intervention (Experimental)
  Interventions: Behavioral: Digital Sensors for Population Awareness about Health Issues using Social Media
- Optimal (Experimental)
  Interventions: Behavioral: Digital Sensors for Population Awareness about Health Issues using Social Media

INTERVENTIONS:
Behavioral: Digital Sensors for Population Awareness about Health Issues using Social Media — A clustered randomized control trial will be conducted and ZIP Codes from each demographic environment will be randomly assigned to control and intervention arms. Digital educational materials about organ donation will be exposed to online users in social media belonging to ZIP Codes assigned to the intervention arm

SUMMARY:
The overarching hypothesis of our study is that social network interventions using artificial intelligence and social media can be used to increase population awareness about health issues. The overarching objective is to improve population awareness on multiple relevant health issues using social network interventions (SNI) and estimate the effect by conducting randomized control trials. Increase population awareness about organ donation in California, especially among minorities

DETAILED DESCRIPTION:
The population of California will be stratified into demographic environments which are groups of ZIP Codes of similar cultural, socioeconomic, and ethnic/racial factors. Digital markers of population awareness about organ donation will be estimated from publicly available online conversations of users in social media. A clustered randomized control trial will be conducted and ZIP Codes from each demographic environment will be randomly assigned to control and intervention arms. Digital educational materials about organ donation will be exposed to online users in social media belonging to ZIP Codes assigned to the intervention arm.

ELIGIBILITY:
Inclusion Criteria:

* Have a California zip code.
* Be a Facebook user

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000000 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change the number of organ donor registration | 3 years
  Measures: number of registrations at Donate Life web page.

SECONDARY OUTCOMES:
Change population awareness about health issues | 3 years
  Measures: number of clicks and impressions on the ad.

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rocha P, Pinheiro D, de Paula Monteiro R, Tubert E, Romero E, Bastos-Filho C, Nuno M, Cadeiras M. Adaptive Content Tuning of Social Network Digital Health Interventions Using Control Systems Engineering for Precision Public Health: Cluster Randomized Controlled Trial. J Med Internet Res. 2023 May 31;25:e43132. doi: 10.2196/43132. PMID 37256680